CLINICAL TRIAL: NCT01327287
Title: Early Aggressive Pain Management is Associated With Improved Outcomes in Blunt Thoracic Trauma
Acronym: Thoracic
Status: Terminated | Type: Observational
Why Stopped: inability to recruit participants despite numerous attempts
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: H9025-35075-01; 10-04955 (Other: UCSF CHR)
Record Dates: First submitted 2011-03-29; First posted 2011-04-01 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Thoracic Injury; Rib Fracture; Sternal Fracture
Keywords: thoracic epidural; blunt; blunt thoracic injury
MeSH Terms: conditions — Thoracic Injuries; Rib Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Trauma patients eligible to receive thoracic epidural: Patients admitted to the hospital suffering from blunt thoracic injury and who meet inclusion/exclusion criteria and receive thoracic epidural for pain
- Control Arm: Trauma patients eligible to receive thoracic epidural but did not receive thoracic epidural for pain

SUMMARY:
This study is designed to analyze the use of early aggressive pain management with thoracic epidural in eligible patients with blunt thoracic trauma.

DETAILED DESCRIPTION:
Due the limited availability of patient population this study requires together with the inclusion and exclusion criteria the study demands, this study will employ both a retrospective chart review process as well as prospective enrollment of qualified patients who provide consent to participate.

The two main groups being evaluated are: (1) eligible patients who received thoracic epidural within 48 hours of injury and (2) eligible patients who did not receive thoracic epidural within 48 hours of injury. In both retrospective and prospective approaches, the investigators will identify patients with blunt thoracic trauma who were eligible for thoracic epidural placement and received the treatment as well as those patients who were eligible but did not receive it. Hospital data such as ventilator days, ICU days, hospital days, hospital charges, and complications, etc. will be recorded.

A retrospective chart review of patients admitted to SFGH suffering from a blunt thoracic injury resulting in 3 or more rib fractures during a 5year time period from January 1, 2004 through January 1, 2009 will be conducted. Patient charts will be reviewed for pain management used for blunt thoracic trauma, hospital course, vitals, labs, and outcome measures. Similar to the prospective enrollment process, the retrospective chart review will screen for patients who had met the inclusion criteria and had not met any exclusion criteria.

Prospective patients admitted to SFGH suffering blunt thoracic injury (rib fractures, sternal fractures) requiring IV opioids for pain relief who do not fit exclusion criteria will be enrolled. Patients will be asked to give informed signed consent for the study doctor to place a thoracic epidural within 48 hours of injury and continued for a maximum of 5 days. The consent process will be twofold. For those who have consented to receive thoracic epidural and agreed to have their health information (HIPAA form) used for the study no additional permission will be required. However, for those patients who do not wish to receive epidural, consent will still be sought if their health information can be used to analyze that arm of the study that did not receive thoracic epidural.

Patient data such as vitals, labs and outcome measures will be recorded and analyzed. The data gathered both in the retrospective and prospective analyses will be used to assess utilization rate of thoracic epidural, and to determine if the use of thoracic epidural is associated with lower resource utilization and is cost effective. In both the retrospective chart review and prospective enrollment process, subjective pain, improved pulmonary function, amount of analgesia and overall clinical outcomes will be measured to determine if patients who received epidural catheters have significantly improved clinical outcomes than those patients who did not receive epidural catheter.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Patients admitted to SFGH trauma service with blunt thoracic trauma (i.e. rib fractures, sternal fractures) requiring IV opioids for pain relief.

Exclusion Criteria:

* Acute spine fractures or pre-existing spine deformity
* Traumatic brain injury or spinal cord injury or altered mental status
* Unstable pelvic fracture or open abdomen
* Hemodynamic instability or major aortic injury (dissection, pseudoaneurysm)
* Coagulopathy
* Mechanical intubation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients > 18 years of age admitted to San Francisco General Hospital Trauma service with blunt thoracic trauma requiring IV opioids for pain relief
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2010-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Hospital Length of stay | An average of 8 weeks
  the hospital length of stay will be assessed for patients who received thoracic epidural compared to those who did not receive thoracic epidural.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco at San Francisco General Hospital, San Francisco, California, United States